CLINICAL TRIAL: NCT06892223
Title: Phase II Clinical Trial to Optimize the Dose of an Anti-NKG2A Monoclonal Antibody (humZ270 MAb, IPH2201) for Patients with Acute Myeloid Leukemia or Myelodysplastic Syndrome Undergoing Haploidentical Transplantation with Post- Transplantation Cyclophosphamide
Brief Title: Anti-NKG2A Monoclonal Antibody for AML or MDS Patients Undergoing Haploidentical Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2020-001; 2024-516974-31-00 (EU CTIS Number); 2020-005902-24 (EudraCT Number)
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukaemia; MDS (Myelodysplastic Syndrome); MPN (Myeloproliferative Neoplasms)
Keywords: MONALIZUMAB; ALLOGENIC TRANSPLANT; ACUTE MYELOID LEUKEMIA; MYELODYSPLASTIC SYNDROM; MYELOPROLIFERATIVE NEOPLASM; GVHD
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders | interventions — monalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- monalizumab treatment arm (Experimental): This study includes a single arm, where all patients will receive Monalizumab (humZ270 mAb, IPH2201), an anti-NKG2A monoclonal antibody, as the intervention. Monalizumab is administered intravenously at a dose of 1 mg/kg on day +30 and day +44 after undergoing haploidentical stem cell transplantation (Haplo-SCT). The use of post-transplantation cyclophosphamide (PT-Cy) is part of the conditioning regimen and inclusion criteria but is not part of the protocol-specified intervention.
  Monalizumab aims to enhance the immune function of NK cells by blocking the NKG2A receptor, potentially improving graft-versus-host disease (GVHD)-free and progression-free survival (GPFS).
  Interventions: Drug: Monalizumab (anti-NKG2A monoclonal antibody)

INTERVENTIONS:
Drug: Monalizumab (anti-NKG2A monoclonal antibody) — Monalizumab (humZ270 mAb, IPH2201) is a humanized IgG4 monoclonal antibody targeting the NKG2A receptor on NK cells. Administered intravenously at a dose of 1 mg/kg on days +30 and +44 after haploidentical stem cell transplantation with post-transplant cyclophosphamide (PT-Cy) as GVHD prophylaxis, Monalizumab aims to enhance NK cell activity by blocking NKG2A. This intervention is unique in its timing, as it is given during a period when CD94/NKG2A+ NK cells are abundant, and its two-dose regimen is designed to optimize NK cell reconstitution. It targets patients with hematologic malignancies, such as AML and MDS, to improve GVHD-free and progression-free survival by enhancing NK cell-mediated immunity. This approach differs from other therapies by focusing on NK cell alloreactivity in the post-transplant setting. Cyclophosphamide is used as part of the pre-transplant conditioning regimen and is part of the inclusion criteria, but it is not part of the protocol-specific intervention.
  Other Names: humZ270; mAb IPH2201

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of the anti-NKG2A monoclonal antibody (Monalizumab) in patients undergoing haploidentical stem cell transplantation (Haplo-SCT) with post-transplantation cyclophosphamide (PT-Cy). The main questions this trial aims to answer are:

* Does Monalizumab improve graft-versus-host disease-free and progression-free survival (GPFS) in patients after Haplo-SCT?
* What are the safety and side effects of Monalizumab in this patient group?
* How does Monalizumab affect the reconstitution and function of NK cells in patients undergoing Haplo-SCT?
* Researchers will administer Monalizumab to participants on day +30 and +44 after transplantation to see if it enhances immune responses and prevents disease relapse or GVHD.

Participants will:

* Receive Monalizumab intravenously at 1 mg/kg on day +30 and day +44 after Haplo-SCT
* Be monitored for clinical outcomes such as GVHD, survival rates, and immune function for up to one year after the transplant
* Undergo regular checkups and tests to assess the effectiveness and safety of the treatment

DETAILED DESCRIPTION:
This Phase II non-randomized, open-label, single-arm, monocentric clinical trial aims to evaluate the safety, efficacy, and biological impact of Monalizumab (humZ270 mAb, IPH2201), an anti-NKG2A monoclonal antibody, in patients undergoing haploidentical stem cell transplantation (Haplo-SCT) with post-transplantation cyclophosphamide (PT-Cy). The study is designed to investigate how the optimization of the dose of this novel antibody can improve the graft-versus-host disease (GVHD)-free and progression-free survival (GPFS) in patients with hematological malignancies, specifically Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS).

Background and Rationale:

Haploidentical stem cell transplantation with PT-Cy as GVHD prophylaxis is a widely used option for patients requiring allogeneic transplantation. However, relapse and GVHD remain significant issues, leading to a GPFS of approximately 30-40%. Alloreactive natural killer (NK) cells play a critical role in graft-versus-tumor (GVT) effects, anti-GVHD, and anti-infectious responses. CD94/NKG2A+ NK cells are prominent early post-transplant, but their effectiveness can be limited. By using anti-NKG2A antibody, NK cell alloreactivity can be enhanced, circumventing the need for an NK alloreactive donor. Preclinical studies have demonstrated that anti-NKG2A antibody treatment restores NK cell-mediated lysis of AML cells, both in vitro and in vivo. This trial aims to assess the clinical benefits of optimizing the dose of anti-NKG2A monoclonal antibody in the Haplo-SCT setting.

Monalizumab is a first-in-class humanized IgG4 antibody targeting the NKG2A receptor on NK cells. It has previously been tested in Phase I trials in solid tumors with promising results at a dosage of 10 mg/kg. In this study, the aim is to optimize the dosage for patients undergoing Haplo-SCT.

Study Design:

This is a non-profit, prospective, open-label, single-arm, monocentric study. The study duration is 5 years, during which participants will receive Monalizumab intravenously at a dose of 1 mg/kg on days +30 and +44 after transplantation. Day +30 is chosen as the starting point for antibody administration as CD94/NKG2A+ NK cells predominate at this time post-transplantation. Additionally, the half-life of Monalizumab is 21 days, meaning two infusions will cover the entire period of NK cell expansion.

The study aims to determine whether the administration of Monalizumab at this timepoint can enhance NK cell alloreactivity and reduce the incidence of GVHD and relapse. The treatment will be stopped if at least three patients develop grade 3-4 acute GVHD after receiving Monalizumab or if any severe adverse events (SAEs) occur that warrant stopping the infusion.

Treatment Plan:

Eligible participants will receive Monalizumab at 1 mg/kg intravenously on days +30 and +44 after undergoing Haplo-SCT. The treatment will be administered as part of the standard care for patients undergoing Haplo-SCT with PT-Cy prophylaxis, which includes Cyclophosphamide (40-50 mg/kg/day on days +3 and +4), Cyclosporine A (3 mg/kg/day starting from day +5), and Mycophenolate Mofetil (45 mg/kg/day from day +5 to day +35).

Primary Objective:

The primary objective of this study is to evaluate the efficacy and safety of Monalizumab in patients undergoing Haplo-SCT with PT-Cy. The primary endpoint is the graft-versus-host disease-free and progression-free survival (GPFS) at one year post-transplantation. This measure will help determine whether Monalizumab improves the overall outcome of patients receiving Haplo-SCT.

Secondary Objectives:

The secondary objectives of this study are:

To evaluate the effect of Monalizumab on the immunological reconstitution of NK cells and other immune cells.

To assess the clinical parameters of survival, toxicity, and the incidence of complications such as relapse, GVHD (both acute and chronic), and post-transplant viral infections.

Endpoints:

Primary Endpoint: The GPFS at 1 year after Haplo-SCT.

Secondary Endpoints:

Clinical Endpoints: Incidence of overall survival (OS), progression-free survival (PFS), non-relapse mortality (NRM), and post-transplant viral infections (including Cytomegalovirus).

Biological Endpoints: Evaluation of NK cell reconstitution and alloreactive functions against leukemic cells following administration of Monalizumab.

Statistical Analysis:

A detailed statistical analysis plan will be followed to address the primary and secondary objectives. Statistical techniques such as Kaplan-Meier analysis will be used to assess survival outcomes, while Cox proportional hazards models will help evaluate the effect of Monalizumab on various clinical and biological parameters. The analysis will include data from all evaluable patients and will be conducted at predefined time points, primarily focusing on the one-year follow-up.

Patient Population:

This study will include adult patients (≥18 years old) with hematologic malignancies, including AML, MDS, and MDS/MPN, who are undergoing Haplo-SCT with PT-Cy. The inclusion criteria are as follows:

Patients capable of providing informed consent and willing to comply with study procedures.

Patients with no HLA-matched donor but who are receiving Haplo-SCT with GVHD prophylaxis.

Patients must have received a myeloablative, reduced intensity, or non-myeloblative conditioning regimen, followed by a bone marrow or peripheral blood stem cell (PBSC) graft.

Women of childbearing potential must use effective contraception during the study.

Safety and Monitoring:

The study will include continuous monitoring for adverse events (AEs) and serious adverse events (SAEs). The occurrence of grade 3-4 acute GVHD following Monalizumab administration will trigger the suspension of the treatment. Regular laboratory tests, physical exams, and imaging (if applicable) will be performed throughout the study to assess the health status of participants. A Data Safety Monitoring Board (DSMB) will oversee the trial to ensure patient safety.

Quality Assurance Plan:

The study will adhere to high standards for data validation and monitoring. Data will be regularly checked for consistency and accuracy against predefined rules. Source data verification will be carried out to ensure that data entered into the study database is complete and accurate. The study will also follow strict SOPs to ensure proper data collection, management, and analysis. Audits will be conducted periodically to ensure compliance with the protocol and regulatory requirements.

Sample Size and Statistical Power:

The sample size for this study has been calculated to provide adequate statistical power (90%) to detect a meaningful difference in GPFS. The goal is to enroll approximately 18 evaluable patients, with a planned interim analysis after the first few patients have completed one year of follow-up.

Plan for Missing Data:

Missing data will be handled using standard statistical techniques such as imputation for missing values, and sensitivity analyses will be performed to account for missing data in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients capable of providing informed consent according to ICH/ GCP, and national/local regulations and be willing to comply with all study-related procedures.
2. Adult patients aged ≥18 years old, without any restriction of gender and race.
3. Patients with a hematologic malignancy represented either by Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) or Myelodysplastic syndrome/Myeloproliferative neoplasm (MDS/MPN).
4. Patients lacking a HLA identical donor and receiving haploidentical stem cell transplant with GVHD/HVG prophylaxis consisting of Cyclophosphamide: 40 or 50 mg/kg/day, day +3 and +4, Cyclosporine A: 3 mg/kg/day from day +5, Mycophenolate mofetil: 45 mg/kg/day, from day +5 to day +35.
5. Patient who has received haplo-SCT with a myeloablative or reduced intensity or nonmyeloblative conditioning followed, either by a bone marrow or a peripheral blood stem cell (PBSC) graft.
6. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test within 8 days prior to start of study drug for women of childbearing potential.
7. Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 52 weeks after the last dose of study therapy. Men with female partners who are of childbearing potential must agree that they will use a highly effective method of contraception from the time of giving informed consent until at least 52 weeks after the patient receives his last dose of study therapy contraception.

Exclusion Criteria:

1. Patients aged < 18 years old.
2. Active uncontrolled infections.
3. CNS involvement of AML disease.
4. Karnofsky performance status (KPS) <60% or severe organ dysfunction, including a left ventricular ejection fraction <40%, DLCO <50% or creatinine clearance <50 ml/min (as per transplant eligibility).
5. Pregnant or breast-feeding or intending to become pregnant during the study.
6. Patients who rapidly relapse after allogenic-SCT before day 30 after allogenic-SCT.
7. Patients who experience acute GVHD before day +30 after allogenic-SCT.
8. Patients treated with a second allogeneic Allo-SCT.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Graft-versus-host disease-free and progression-free survival (GPFS) | GPFS will be evaluated 1 year after Haplo-SCT with PT-Cy and Monalizumab administration on day +30 and +44.
  GPFS is defined as the time from Haplo-SCT with post-transplant cyclophosphamide (PT-Cy) until the occurrence of either graft-versus-host disease (GVHD) or disease progression/relapse. This measure evaluates the combined effect of Monalizumab (NKG2A blockade) in preventing both GVHD and disease progression. It is a comprehensive indicator of treatment efficacy, assessing whether the addition of Monalizumab improves patient outcomes by prolonging the period free of both GVHD and disease progression.

SECONDARY OUTCOMES:
Overall Survival (OS) | Overall Survival (OS) will be evaluated at 1 year after Haplo-SCT
  Overall Survival (OS) is defined as the time from Haplo-SCT with post-transplant cyclophosphamide (PT-Cy) and Monalizumab administration until death from any cause. It is a key indicator of the overall benefit of the treatment, evaluating whether the addition of Monalizumab improves long-term survival in patients undergoing Haplo-SCT.
Progression-Free Survival (PFS) | PFS will be evaluated at 1 year after Haplo-SCT
  Progression-Free Survival (PFS) is defined as the time from Haplo-SCT with post-transplant cyclophosphamide (PT-Cy) and Monalizumab administration until the occurrence of disease progression or relapse. PFS evaluates the efficacy of Monalizumab in delaying or preventing the progression of hematological malignancies, such as Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS), after Haplo-SCT.
Non-Relapse Mortality (NRM) | NRM will be evaluated at 1 year after Haplo-SCT
  Non-Relapse Mortality (NRM) refers to mortality from causes other than disease relapse or progression, such as complications due to GVHD, infections, or other treatment-related toxicities. NRM will evaluate whether Monalizumab affects the risk of death from non-disease related causes in patients post-Haplo-SCT.
Incidence of Acute and Chronic GVHD | GVHD incidence will be assessed at 6 months and 1 year after Haplo-SCT
  This measure tracks the incidence of acute and chronic GVHD in patients after Haplo-SCT with PT-Cy and Monalizumab treatment. It evaluates whether the addition of Monalizumab affects the rate of GVHD development.
Post-transplant Viral Infections | Post-transplant viral infections will be assessed until 100 days after Haplo-SCT
  The incidence of viral infections (such as CMV, EBV, etc.) will be monitored in patients after Haplo-SCT. This measure will evaluate whether Monalizumab influences the incidence of viral infections post-transplant.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale Policlinico San Martino, Genova, GENOVA
  - Irccs Istituto Clinico Humanitas, Rozzano, MILANO

IPD SHARING:
Plan to Share IPD: No